CLINICAL TRIAL: NCT06416696
Title: Toripalimab Combined With Chemoradiotherapy Followed by Toripalimab Maintenance Therapy for High-risk Locally Advanced Cervical Cancer: the Phase II Single-arm TorCH -CC Study
Brief Title: Toripalimab for High-risk Locally Advanced Cervical Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, SHUANG ZHENG JIA, PhD, Attending Physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TorCH-CC
Record Dates: First submitted 2024-05-11; First posted 2024-05-16 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancers
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — toripalimab; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab combined with Chemoradiotherapy followed by Toripalimab maintenance therapy (Experimental): Toripalimab combined with Chemoradiotherapy followed by Toripalimab maintenance therapy for High-risk Locally Advanced Cervical Cancer
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — 1. Radiotherapy: Both external beam and brachytherapy, with radiation therapy techniques, target delineation, prescribed doses, and organ-at-risk constraints following established guidelines.
  2. Chemotherapy: The preferred regimen is cisplatin at a dose of 40mg/m^2 administered intravenously once weekly for 5-6 cycles; for patients intolerant to cisplatin or with renal impairment, carboplatin (AUC=2) may be considered, also administered once weekly.
  3. Toripalimab concurrent immunotherapy: Following the regimens of phase III RCTs such as JUPITER-02, JUPITER-06, CHOICE-01, NEOTORCH, and RENOTORCH, Toripalimab is administered at a fixed dose of 240mg per infusion, given intravenously once every 3 weeks for three doses.
  4. The concurrent chemoradiotherapy and immunotherapy phase does not exceed 8 weeks in duration.
  Other Names: Radiotherapy; Chemotherapy(cisplatin)

SUMMARY:
This phase II clinical study assesses the efficacy and safety of Toripalimab combined with chemoradiotherapy (CRT) followed by Toripalimab maintenance in treating high-risk locally advanced cervical cancer (HR-LACC). Despite CRT being the standard treatment, HR-LACC patients face poor survival outcomes. Toripalimab, a cost-effective PD-1 inhibitor, has shown promise in prior research. The primary endpoint is 2-year progression-free survival, with the study aiming to improve treatment accessibility and patient prognoses in China.

DETAILED DESCRIPTION:
Cervical cancer is the most prevalent malignant tumor of the female reproductive system in China, with an estimated 150,700 new cases and 55,700 new deaths annually. Concurrent chemoradiotherapy (CRT) remains the standard treatment for locally advanced cervical cancer (LACC). However, for high-risk LACC (HR-LACC) patients, the 2-year progression-free survival (PFS) rate is only 57%-62%, and the 5-year overall survival (OS) rate is 52%-64%, which are the leading causes of patient mortality. The KEYNOTE-A18 study demonstrated that the combination of pembrolizumab and CRT reduced the progression risk and death risk by 30% and 27%, respectively, for HR-LACC patients. Following this, the FDA approved pembrolizumab in combination with CRT for the treatment of newly diagnosed stages III-IVA cervical cancer in January 2024. Nevertheless, the high cost of pembrolizumab poses a significant barrier for patients in China. Toripalimab, the first domestically approved PD-1 inhibitor in China, has shown good safety and efficacy in previous studies and is more affordable. This phase II, single-arm, open-label study aims to evaluate the efficacy and safety of Toripalimab combined with CRT followed by Toripalimab maintenance therapy in 130 patients with stages III-IVA cervical cancer. The primary endpoint is the 2-year PFS. The study is expected to contribute to the implementation of precision and personalized treatment for HR-LACC in China, with the potential to improve patient survival rates and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed cervical squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma.
2. FIGO 2018 staging criteria classifying the disease as stages III-IVA.
3. Age range from 18 to 70 years inclusive.
4. No prior receipt of surgery, radiotherapy, or systemic anticancer therapy for the treatment of cervical cancer.
5. No previous exposure to the study drug.
6. Presence of at least one measurable or evaluable lesion as per RECIST version 1.1, with the measurable lesion exhibiting a longest diameter of ≥10 mm on spiral CT scan or a shortest diameter of ≥15 mm for enlarged lymph nodes, which has not been previously irradiated.
7. Absence of central nervous system diseases, both primary and metastatic.
8. WHO/ECOG performance status score of 0-1.
9. Anticipated survival duration of at least 12 weeks.
10. Adequate organ function within the following parameters (without the use of any blood components, cytokines, or growth factors within 14 days prior to randomization):

    1. Absolute neutrophil count (ANC) ≥1.5×10^9/L
    2. Platelet count ≥90×10^9/L
    3. Hemoglobin level ≥90 g/L
    4. Serum albumin level ≥30 g/L
    5. Bilirubin level ≤1.5 times the upper limit of normal (ULN)
    6. Alanine transaminase (ALT) and aspartate transaminase (AST) levels ≤3×ULN
    7. Serum creatinine level ≤1.5×ULN
    8. Thyroid-stimulating hormone (TSH) level ≤1×ULN (with eligibility also extended to patients with free triiodothyronine [FT3] or free thyroxine [FT4] levels ≤1×ULN).
11. For women of childbearing potential not undergoing surgical sterilization, a negative serum pregnancy test (hCG) within 72 hours prior to study randomization is required; breastfeeding must be absent. Additionally, the use of a medically approved contraceptive method is mandatory from the time of informed consent through the study treatment period and for 120 days following the final administration of the trial medication or 180 days after the last chemotherapy/radiotherapy session. Participants must also agree not to donate eggs for reproductive purposes or to freeze/preserve eggs for this use during the aforementioned period.
12. Provision of a tumor tissue biopsy specimen is mandatory.
13. Informed consent must be obtained with documentation.
14. Availability for follow-up assessments.

Exclusion Criteria:

* 1. Known hypersensitivity to any component of the study medication. 2. Participation in other clinical trials, with a washout period of less than 4 weeks following completion.

  3. Prior treatment with immune checkpoint inhibitors, including but not limited to other anti-PD-1 and anti-PD-L1 monoclonal antibodies.

  4. Patients requiring immunosuppressive pharmacotherapy. 5. Individuals requiring systemic or absorbable topical corticosteroids at immunosuppressive doses. Use of prednisone at a dosage greater than 10mg/day or equivalent is prohibited within two weeks of study drug administration.

  6. Presence of active autoimmune diseases or a history thereof, excluding vitiligo, resolved childhood asthma, or resolved atopic diseases. Patients with asthma requiring intermittent bronchodilator therapy or other interventions are also excluded.

  7. Active infectious processes necessitating antimicrobial therapy, including the use of antibacterial, antiviral, or antifungal agents.

  8. History of immunodeficiency, including HIV seropositivity or other acquired and congenital immunodeficiency disorders.

  9. Uncontrolled cardiac symptoms or diseases, such as NYHA class II or higher heart failure, unstable angina, myocardial infarction within the past year, atrial fibrillation, clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention, PR interval greater than 250 ms, or QTc interval ≥470 ms.

  10. A history of arterial or venous thromboembolic events within the past 6 months.

  11. Poorly controlled hypertension despite antihypertensive therapy (systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg).

  12. Proteinuria of 2+ or higher and a 24-hour urinary protein excretion exceeding 1.0 g.

  13. Coagulopathy (INR >2.0, PT >16 seconds), a bleeding diathesis, or concurrent anticoagulation or thrombolytic therapy.

  14. Bilateral hydronephrosis, unless resolved by unilateral stent placement or percutaneous nephrostomy, or deemed mild and without clinical significance by the investigator.

  15. Contraindications to chemotherapy administration. 16. Contraindications to receiving brachytherapy. 17. History of other malignancies within the past 5 years, except for basal cell carcinoma and squamous cell carcinoma of the skin.

  18. Administration of live vaccines within 4 weeks preceding the first dose of the trial medication. Inactivated seasonal influenza vaccines are permissible.

  19. History of substance abuse that has not been successfully managed or presence of psychiatric disorders that may interfere with study participation.

  20. Any medical, psychiatric, or social conditions deemed by the investigator to potentially impact the subject's ability to provide informed consent, participate fully in the study, or affect the interpretability of the study results.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 2 year
  2-year progression-free survival (PFS) rate as assessed by the investigator

SECONDARY OUTCOMES:
short-term efficacy assessment | 30 days (±7 days) and 90 days (±7 days) after the last dose
  ORR Duration of efficacy (DoR)
side effects | 30 days (±7 days) and 90 days (±7 days) after the last dose
  Treatment-related Side Effects (TRAEs) and immune-related Side Effects (iRAEs)
OS | 2 years
  2 years of investigator evaluation -OS and PFS, OS
quality of life assessments | 30 days (±7 days) and 90 days (±7 days) after the last dose
  quality of life assessments utilizing the EORTC QLQ-C30 v3.0

CONTACTS AND LOCATIONS:
Overall Officials: SHUANGZHENG JIA, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No